CLINICAL TRIAL: NCT04602572
Title: Obesity and Oral Diseases in Adult Patients
Acronym: ObOd
Status: Not yet recruiting | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Knut N. Leknes, Professor, University of Bergen
Other Study IDs: 152810
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-04

CONDITIONS: Obesity; Oral Diseases; Periodontitis; Dental Caries; Dental Erosion
Keywords: Obesity; Overweight; Periodontitis; Caries; Bariatric surgery; Oral health
MeSH Terms: conditions — Obesity; Periodontitis; Dental Caries; Tooth Erosion; Overweight | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-surgical group.: Patients will be offered a standardized program comprised of individual consultations by a trained nurse every 3 months over 2 years, participation in a lifestyle course with 13 group sessions focusing on healthy diet and physical activity, and pharmacotherapy.
  Interventions: Behavioral: Lifestyle course.
- Surgical group: After completing the systematic work-up and the lifestyle course, eligible subjects will be offered bariatric surgery. The surgical procedure will be chosen at the surgeon's discretion taking into consideration the target weight, comorbidities, risk of complications, the patient's ability to cope with side effects and complications, and the patient's motivation.
  Interventions: Procedure: Bariatric surgery.

INTERVENTIONS:
Behavioral: Lifestyle course. — Pharmacotherapy
  Groups: Non-surgical group.
Procedure: Bariatric surgery. — Sleeve gastrectomy or gastric bypass.
  Groups: Surgical group

SUMMARY:
Overweight and obesity are among the major chronic disorders of the 21st century and one of the fastest growing health problems worldwide. Obesity is accompanied by a state of low-grade inflammation which may contribute to the occurrence of diabetes mellitus, cardiovascular disease, hypertension, stroke, and certain cancers. Furthermore, obesity has been associated with oral health problems as hyposalivation, dental caries and periodontitis.

The management and treatment of obesity is outlined in clinical guidelines from American Association of Clinical Endocrinologists/American College of Endocrinology and European Association for the Study of Obesity. The cornerstone is life-style modification programs aiming to reduce energy intake and increase physical activity, referred to as conservative treatment. All patients must undergo a thorough systematic work-up. The work-up concludes in a final multi-disciplinary meeting with a concrete individualized plan on how sustained weight-loss is to be achieved; either by a non-surgical or a surgical approach (Bariatric surgery).

Periodontitis is cited to be the sixth most prevalent chronic condition globally. The mechanisms by which obesity affects the periodontal tissues is poorly understood, and the understanding of the key role of adipocytes in the inflammatory response to infections is crucial in comprehending how periodontal disease susceptibility may be modified in obese individuals.

The main objectives of the present research project are to explore the association between obesity and oral diseases and further, to assess how weight changes following non-surgical and surgical interventions of obese patients may affect the cariological and periodontal health status.

Four hundred patients referred to the Obesity Centre at Haukeland University Hospital, Norway will consecutively be screened and invited to participate in this prospective cohort study. At baseline, detailed medical and oral data will be obtained from health forms, questionnaires, clinical examinations, and by consulting the patient's care team. Following baseline examination, all patients will undergo a thorough systematic work-up consisting av interviews and consultations concluding in a final multi-disciplinary individualized non-surgical or surgical treatment plan on how sustained weight-loss can be achieved. New sets of medical, oral, and molecular data will be collected at 3-, 12- and 18-month following non-surgical/surgical interventions.

DETAILED DESCRIPTION:
The management and treatment of obesity is outlined in clinical guidelines from American Association of Clinical Endocrinologists/American College of Endocrinology (AACE/ACE), European Association for the Study of Obesity (EASO) and others. The cornerstone is life-style modification programs aiming to reduce energy intake and increase physical activity, often referred to as conservative treatment. In recent years, pharmacological management to achieve weight loss is increasingly used as effective drugs become available. Conservative treatment generally targets to induce long-term weight loss of 5-10%. The obesity treatment has wider objectives than weight loss alone by also including treatment of obesity-related comorbidities like diabetes mellitus, hypertension, dyslipidemia, and obstructive sleep apnea with the ultimate goals of improving quality of life, working ability and reduce mortality.

Bariatric surgery is considered an effective and safe intervention for the treatment of obesity. Consistent with international consensus gastrointestinal surgery might be recommended for patients with extreme obesity (BMI ≥ 40 kg/m2) as well as for those with BMI ≥ 35 kg/m2 with significant comorbidities. The surgical procedures are usually performed laparoscopically, and includes sleeve gastrectomy, Roux-en-Y gastric bypass and biliopancreatic diversion with duodenal switch.

Benefits of bariatric surgeries include significant weight loss, improved and remission of obesity-related comorbidities such as type 2 diabetes, hyperlipidemia, hypertension, cardiovascular disease, obstructive sleep apnea, anxiety, depression, and improved quality of life. Gastro esophageal reflux and vomiting in addition to increased intake of food and drinks have been reported as potential side effects. All these side effects are considered risk factors for the occurrence of dental caries and dental erosion, which may lead to decreased function and pain. Periodontitis is also reported to be more frequent in individuals who have undergone bariatric surgery probably related to nutritional deficiency secondary to the surgery.

Periodontitis is a widespread chronic, inflammatory disease of the gingival tissues and alveolar bone triggered by oral biofilms. Since 2010, periodontitis is cited to be the sixth most prevalent chronic condition globally. The high prevalence of moderate/severe periodontitis may be attributed to multiple factors such as lifestyle, genetics, and medical care. Current knowledge recognizes adipose tissue as an endocrine organ in which adipocytes play an important role as inflammatory modulators, producing anti- and pro-inflammatory cytokines which regulate oral and systemic inflammation. In obese individuals, an imbalance may result in an increased expression of pro-inflammatory and reduction of anti-inflammatory adipokines, leading to the establishment of a chronic inflammatory status.

Available data on obesity and oral diseases as well as the influence of non-surgical and surgical interventions on oral health are scarce, and several reports have published conflicting and inconsistent results. The main objectives of the present research project are to explore the association between obesity and oral diseases and assess how weight changes following non-surgical and surgical interventions may affect the cariological and periodontal health status.

Pre-study protocols and tests. This cohort study will enroll patients in need for obesity therapy at Haukeland University Hospital, Bergen, Norway. The study protocol and informed consent, following the Helsinki Declaration of 1975, version 2008, has been submitted to the Medical Research Ethics Committee, University of Bergen, Norway (reference 152810). Each patient will read and sign the informed consent prior to inclusion in the study.

Study subjects. Patients referred to the Obesity Centre at Haukeland University Hospital will consecutively be screened for eligibility from January 2021 through December 2021. Four hundred patients will be invited to participate in this prospective cohort study. At baseline, detailed medical and oral data will be obtained from health forms, questionnaires, clinical examinations (including weight and height registrations), and by consulting the patient's care team. Following baseline examination/registration, the patients will be allocated either to non-surgical or surgical interventions according to established medical guidelines. At 3-month control post-surgery, periodontal and cariological clinical data together with local and systemic molecular data will be obtained from each patient. The follow-up controls at 12 and 18 months will contain a complete set of data collection including medical, dental, and molecular parameters.

Treatment. All patients will undergo a thorough systematic work-up. The first interview will be conducted by a trained nurse. Data regarding social and occupational situation, social network, daily activity levels, weight history, personal resources, and barriers to achieve sustained weight loss will be collected. The second consultation will be done by a physician, focusing on identifying and optimizing medical and psychiatric disorders. The third interview will be done by clinical nutritionist to assess eating habits. If needed, the patient will also be evaluated by a physiotherapist, psychologist and/or be referred to further investigations at the respiratory, cardiac, and orthopedic departments. The work-up concludes in a final multi-disciplinary meeting with a concrete individualized plan on how sustained weight-loss is to be achieved.

Non-surgery group. In this group, included patients will be offered a standardized program comprised of individual consultations by a trained nurse every 3 months over 2 years. Furthermore, they will participate in a lifestyle course with 13 group sessions focusing on healthy diet and activity based on the recommendations of the Norwegian Directorate of Health. Other therapeutic options include pharmacotherapy to reduce weight (GLP1 analogues or naltrekson/bupropion) as well as treatment of comorbidities (diabetes mellitus, hypertension, dyslipidemia, sleep-apnea, etc.).

Surgery group. After completing the systematic work-up and the lifestyle course, eligible subjects will be offered bariatric surgery. The surgical procedure will be chosen at the surgeon's discretion taking into consideration the target weight, comorbidities, risk of complications, the patient's ability to cope with side effects and complications, and the patient's motivation. Generally, sleeve gastrectomy has lower incidence of severe side effects compared with gastric bypass (Roux-en-Y gastric bypass) or mini-bypass but are less effective in terms of weight loss and amelioration of obesity-related comorbidities. After surgery, patients will be followed up at the outpatient clinic 2, 12, 24 months and 5 and 10 years postoperatively.

Periodontal diagnosis. Periodontitis will be diagnosed by using the criteria of World Workshop on the Classification of Periodontal and Peri-implant Diseases and Conditions.

Smoking status. Smoking status will be registered as current, former, or never smoker. Self-reported smoking experience will be calculated in pack years; the number of cigarettes smoked daily multiplied by the number of years divided by 20 (a standard pack of cigarettes). In addition, smoking status will be objectively validated by measuring cotinine levels in serum.

Medical examination. Data about current medications, past medical history including cardiovascular events, arterial hypertension, BMI, waist-to-hip ratio (WHR) and smoking habit will be collected. Glycated hemoglobin (HbA1c) will be measured by standard laboratory methods, whereas high-sensitivity C reactive protein (CRP) will be determined in serum by particle-enhanced immune-nephelometry (hsCRP kit, Dade Behring, Eschborn, Germany).

Oral radiographs, and clinical periodontal and cariological examination. Before clinical examination, a full mouth series of intraoral radiographs will be taken. The following periodontal parameters will be registered at baseline and at 3, 12 and 18 months: PD as the distance in mm from the gingival margin to the probable base of the pocket at six sites; CAL as the distance in mm from the cementoenamel junction (CEJ) to the probable base of the pocket at six sites (PCP, UNC 15, Hu-Friedy, Chicago, IL, USA); full mouth dental plaque scores recorded as the percentage of tooth surfaces with visible plaque at the mesial, distal, buccal and lingual surfaces following staining with disclosing solution; full mouth bleeding on probing (BoP) as the presence of bleeding after gentle probing.

A full mouth cariological examination including dental caries and dental erosion will be performed for the non-surgical and surgical group at baseline and at 12 and 18 months after bariatric surgery (matching timepoints for both groups). This will include radiographs (bitewings), intraoral photos and cast models made from tooth impressions. In combination with established indexes, these data will provide reliable measurements of the cariological disease status.

Gingival crevicular fluid assessments and saliva analysis. Sample sites will be isolated with cottons rolls, carefully cleaned for supragingival plaque and air-dried. A perio paper strip will then be gently placed one to two mm into the entrance of the pocket and left in place for 30 seconds. For quantitative measurements, the perio paper will be inserted into the Periotron 8000® (Oraflow Inc, Smithtown, NY, USA), a previously calibrated instrument to measure the volume of fluid collected. Gingival crevicular fluid (GCF) volume will be measured at baseline and at 3, 12 and 18 months. Strips will be immediately inserted into separate and dry microtubes, labelled, and stored at 80°C until further analysis.

Unstimulated salivary samples (5 mL) will be collected from each patient between 8 am and 10 am. The patients will rinse their mouth with water 5 minutes before sample collection. The first saliva expectoration will be discarded to avoid food and any other substances capable of contaminating the sample to interfere with the results of the biochemical analyses. The patients will also be instructed to refrain from brushing their teeth and eating or drinking 60 minutes before sample collection.

In addition, pH of both unstimulated and paraffin-stimulated saliva samples will be measured, and a small aliquot of the stimulated saliva will be used to determine the buffer capacity. Saliva samplings and qualitative and quantitative analyzes will be performed at baseline and at 3, 12 and, 18 months follow-ups for both groups.

Questionnaire. At baseline, a questionnaire including 27 multiple-choice questions will be distributed to the participants.

Statistical analysis. The sociodemographic data of the patients will be described using descriptive statistics. Age, BMI, medical and oral parameters, and the amount of analyzed local and systemic biomarkers will be expressed as median and inter-quartile range (IQR). For the cross-sectional analysis, linear regression models and logistic regression models will be used to adjust for potential confounding factors. For analysis of differences over time between groups (e.g. operated versus non-operated patients) generalized estimation equations (linear and logistic models) will be performed, adjusting for potential confounding factors. Furthermore, as a causal approach, homogenous groups will be compared using propensity matched samples. The standard approach using regression models and the propensity score matching will furthermore be compared with analysis using inverse probability weighted models. Differences and changes will be considered significant with a two-sided p-value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Obese adult patients.
* Patients referred to the Obesity Clinic at the Hospital.

Exclusion Criteria:

* Unwillingness to participate.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese adults referred to the Obesity Centre from primary, secondary, and tertiary health services.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in probing depth (PD) | 18 months.
  PD: The vertical distance from the gingival margin to the probable base of the pocket in mm.
Change in clinical attachment level (CAL) | 18 months.
  CAL: The vertical distance from the cemento-enamel junction or the margin of a dental restoration to the probable base of the pocket in mm.

SECONDARY OUTCOMES:
Bleeding on probing (BoP). | 18 months.
  At site level, BoP will be recorded as present upon gentle probing to the base of the pocket.
Gingival crevicular fluid (GCF). | 18 months.
  Sites will be isolated with cottons rolls, cleaned for supragingival plaque, and air-dried. A perio paper strip will then be placed 1-2 mm into the orifice of the site and left in place for 30 sec. The perio strip will be inserted into the Periotron 8000® (Oraflow, Smithtown, NY, USA) calibrated to estimate the volume of GCF collected.
Unstimulated saliva. | 18 months.
  Salivary collection will be performed directly into a sterile tube (Epperdorf North America, Hauppauge, NY).
Whole blood | 18 months.
  A volume of 5 ml peripheral blood will be obtained from each patient by venipuncture in the antecubital fossa following an overnight fast.
Tooth loss | 18 months
  The number of missing teeth will be counted at baseline and after 18 months observation.
Dental caries | 18 months
  Caries will be quantitatively scored according to Espelid & Tveits clinical index based on six (6) grades (0-5) where 0 indicates no caries and 5 deep caries into the inner third of dentin. Caries will be scored at baseline and at 18 months.
Dental erosion | 18 months
  Dental erosion will be quantitatively scored according to the VEDE clinical index system based on six (6) grades (0-5) where 0 indicates no erosion and 5 > 2/3 of the surface exposed. Dental erosion will be scored at baseline and at 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Knut N Leknes, Professor, Principal Investigator — Bergen5032#

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marsicano JA, Sales-Peres A, Ceneviva R, de C Sales-Peres SH. Evaluation of oral health status and salivary flow rate in obese patients after bariatric surgery. Eur J Dent. 2012 Apr;6(2):191-7. PMID 22509123
- [Background] Garvey WT, Mechanick JI, Brett EM, Garber AJ, Hurley DL, Jastreboff AM, Nadolsky K, Pessah-Pollack R, Plodkowski R; Reviewers of the AACE/ACE Obesity Clinical Practice Guidelines. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY COMPREHENSIVE CLINICAL PRACTICE GUIDELINES FOR MEDICAL CARE OF PATIENTS WITH OBESITY. Endocr Pract. 2016 Jul;22 Suppl 3:1-203. doi: 10.4158/EP161365.GL. Epub 2016 May 24. PMID 27219496
- [Background] Yumuk V, Tsigos C, Fried M, Schindler K, Busetto L, Micic D, Toplak H; Obesity Management Task Force of the European Association for the Study of Obesity. European Guidelines for Obesity Management in Adults. Obes Facts. 2015;8(6):402-24. doi: 10.1159/000442721. Epub 2015 Dec 5. PMID 26641646
- [Background] Apovian CM, Aronne LJ, Bessesen DH, McDonnell ME, Murad MH, Pagotto U, Ryan DH, Still CD; Endocrine Society. Pharmacological management of obesity: an endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2015 Feb;100(2):342-62. doi: 10.1210/jc.2014-3415. Epub 2015 Jan 15. PMID 25590212
- [Background] Barbosa CS, Barberio GS, Marques VR, Baldo Vde O, Buzalaf MA, Magalhaes AC. Dental manifestations in bariatric patients: review of literature. J Appl Oral Sci. 2009;17 Suppl(spe):1-4. doi: 10.1590/s1678-77572009000700002. PMID 21499648
- [Background] Costa RC, Yamaguchi N, Santo MA, Riccioppo D, Pinto-Junior PE. Outcomes on quality of life, weight loss, and comorbidities after Roux-en-Y gastric bypass. Arq Gastroenterol. 2014 Jul-Sep;51(3):165-70. doi: 10.1590/s0004-28032014000300002. PMID 25296074
- [Background] Mechanick JI, Youdim A, Jones DB, Garvey WT, Hurley DL, McMahon MM, Heinberg LJ, Kushner R, Adams TD, Shikora S, Dixon JB, Brethauer S; American Association of Clinical Endocrinologists; Obesity Society; American Society for Metabolic & Bariatric Surgery. Clinical practice guidelines for the perioperative nutritional, metabolic, and nonsurgical support of the bariatric surgery patient--2013 update: cosponsored by American Association of Clinical Endocrinologists, The Obesity Society, and American Society for Metabolic & Bariatric Surgery. Obesity (Silver Spring). 2013 Mar;21 Suppl 1(0 1):S1-27. doi: 10.1002/oby.20461. PMID 23529939
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Poirier P, Cornier MA, Mazzone T, Stiles S, Cummings S, Klein S, McCullough PA, Ren Fielding C, Franklin BA; American Heart Association Obesity Committee of the Council on Nutrition, Physical Activity, and Metabolism. Bariatric surgery and cardiovascular risk factors: a scientific statement from the American Heart Association. Circulation. 2011 Apr 19;123(15):1683-701. doi: 10.1161/CIR.0b013e3182149099. Epub 2011 Mar 14. No abstract available. PMID 21403092
- [Background] Basoglu OK, Vardar R, Tasbakan MS, Ucar ZZ, Ayik S, Kose T, Bor S. Obstructive sleep apnea syndrome and gastroesophageal reflux disease: the importance of obesity and gender. Sleep Breath. 2015 May;19(2):585-92. doi: 10.1007/s11325-014-1051-4. Epub 2014 Aug 31. PMID 25173794
- [Background] Jastrzebska-Mierzynska M, Ostrowska L, Wasiluk D, Konarzewska-Duchnowska E. Dietetic recommendations after bariatric procedures in the light of the new guidelines regarding metabolic and bariatric surgery. Rocz Panstw Zakl Hig. 2015;66(1):13-9. PMID 25813068
- [Background] Netto BD, Moreira EA, Patino JS, Beninca JP, Jordao AA, Frode TS. Influence of Roux-en-Y gastric bypass surgery on vitamin C, myeloperoxidase, and oral clinical manifestations: a 2-year follow-up study. Nutr Clin Pract. 2012 Feb;27(1):114-21. doi: 10.1177/0884533611431462. PMID 22307495
- [Background] de Moura-Grec PG, Yamashita JM, Marsicano JA, Ceneviva R, de Souza Leite CV, de Brito GB, Brienze SL, de Carvalho Sales-Peres SH. Impact of bariatric surgery on oral health conditions: 6-months cohort study. Int Dent J. 2014 Jun;64(3):144-9. doi: 10.1111/idj.12090. Epub 2014 Jan 11. PMID 24410073
- [Background] Meyle J, Chapple I. Molecular aspects of the pathogenesis of periodontitis. Periodontol 2000. 2015 Oct;69(1):7-17. doi: 10.1111/prd.12104. PMID 26252398
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Trends in adult body-mass index in 200 countries from 1975 to 2014: a pooled analysis of 1698 population-based measurement studies with 19.2 million participants. Lancet. 2016 Apr 2;387(10026):1377-1396. doi: 10.1016/S0140-6736(16)30054-X. PMID 27115820
- [Background] Dye BA. Global periodontal disease epidemiology. Periodontol 2000. 2012 Feb;58(1):10-25. doi: 10.1111/j.1600-0757.2011.00413.x. No abstract available. PMID 22133364
- [Background] Karlsson L, Carlsson J, Jenneborg K, Kjaeldgaard M. Perceived oral health in patients after bariatric surgery using oral health-related quality of life measures. Clin Exp Dent Res. 2018 Oct 16;4(6):230-240. doi: 10.1002/cre2.134. eCollection 2018 Dec. PMID 30603104
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- [Background] Scott DA, Palmer RM, Stapleton JA. Validation of smoking status in clinical research into inflammatory periodontal disease. J Clin Periodontol. 2001 Aug;28(8):715-22. doi: 10.1034/j.1600-051x.2001.280801.x. English, French, German. PMID 11442730
- [Background] Barros SP, Williams R, Offenbacher S, Morelli T. Gingival crevicular fluid as a source of biomarkers for periodontitis. Periodontol 2000. 2016 Feb;70(1):53-64. doi: 10.1111/prd.12107. PMID 26662482
- [Background] Bunaes DF, Mustafa M, Mohamed HG, Lie SA, Leknes KN. The effect of smoking on inflammatory and bone remodeling markers in gingival crevicular fluid and subgingival microbiota following periodontal therapy. J Periodontal Res. 2017 Aug;52(4):713-724. doi: 10.1111/jre.12438. Epub 2017 Mar 17. PMID 28306142
- [Derived] Nilsen A, Thorsnes A, Lie SA, Methlie P, Bunaes DF, Reinholtsen KK, Leknes KN. Periodontitis in obese adults with and without metabolic syndrome: a cross-sectional study. BMC Oral Health. 2023 Jul 1;23(1):439. doi: 10.1186/s12903-023-03133-5. PMID 37393272